CLINICAL TRIAL: NCT04732312
Title: Impact of Formal Home Help on Quality of Life for Caregivers of Elderly Patients With Neurocognitive Impairment: a Prospective Monocenter Study
Brief Title: Impact of Formal Home Help on Quality of Life for Caregivers of Elderly Patients With Neurocognitive Impairment
Acronym: PIAF-QVA
Status: Terminated | Type: Observational
Why Stopped: recruitment issues
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Other Study IDs: GHRMSA 952; ID-RCB 2018-A02307-48 (Other: ANSM)
Record Dates: First submitted 2021-01-14; First posted 2021-02-01 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2018-11

CONDITIONS: Age-related Cognitive Decline
Keywords: cognitive impairment; caregiver quality of life; caregiver burden; caregiver vulnerability
MeSH Terms: conditions — Cognitive Dysfunction; Caregiver Burden

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Home help — Setting up of a formal home help

SUMMARY:
The purpose of this prospective monocenter observational study is to assess the impact of the first introduction of formal home help (personalized autonomy allowance for seniors) on the quality of life of home caregivers of elderly patients with neurocognitive impairment.

DETAILED DESCRIPTION:
An aging population is leading to an increase in neurodegenerative disorders that are responsible for loss of autonomy. In order to keep patients with neurocognitive impairment at home, the availability of home caregivers is essential. The neurocognitive deterioration of elderly patients is a significant burden for home caregivers and can affect their quality of life. The implementation of formal home help (personalized autonomy allowance for seniors) can relieve home caregivers and improve their quality of life.

Conduct of research:

Elderly patients followed in the geriatric department of the Mulhouse French hospital, and for whom a formal home help (personalized autonomy allowance for seniors) is initiated will be recruited. The evolution of home caregiver's quality of life, burden and vulnerability, will be assessed during three months.

ELIGIBILITY:
Inclusion criteria:

* Patient 60 years of age or older
* Diagnosis of neurocognitive disorders
* MMSE score less than or equal to 26
* GIR score inferior or equal to 4
* Introduction of formal home help (personalized autonomy allowance for seniors program)
* Patient living in Haut-Rhin department (France)
* Patient receiving regular informal help at home (at least once a week)
* Availability of the current home helper to participate in the sudy
* Non-opposition to participation in the study

Exclusion criteria:

* Introduction of formal home care not related to the personalized autonomy allowance program
* Patient under legal protection

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elderly people with neurocognitive disorders benefiting from a home support program (personalized autonomy allowance for seniors program).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Caregiver quality of life | 90 days
  Variation of caregiver quality of life between inclusion and 90 days. Quality of life is assessed with the PIXEL study evaluation scale. This is a 20-item scale, subdivided in four domains: behavioral capacities to face difﬁculties generated by the patient, relation with the environment, psychological perception of the situation, perception of a possible distress. Score ranges from 0 to 100 points (5 points for each item).

SECONDARY OUTCOMES:
Caregiver vulnerability | 90 days
  Variation of caregiver vulnerability between inclusion and 90 days. Vulnerability is assessed through another PIXEL study 20-item evaluation scale. Score ranges from 0 to 100 points.
Caregiver burden | 90 days
  Variation of caregiver burden between inclusion and 90 days. Burden is assessed with the 7-item mini-Zarit scale. Score ranges from 0 to 7.
Caregiver quality of life according to the type of formal home care | 90 days
  Variation of caregiver quality of life between inclusion and 90 days. Quality of life is assessed with the PIXEL study evaluation scale.
Caregiver vulnerability according to the type of formal home care | 90 days
  Vulnerability is assessed through another PIXEL study 20-item evaluation scale.
Caregiver burden according to the type of formal home care | 90 days
  Variation of caregiver burden between inclusion and 90 days. Burden is assessed with the 7-item mini-Zarit scale. Score ranges from 0 to 7.
Variation of quality of life score according to each domain | 90 days
  Evolution of quality of life according to each domain of the PIXEL study evaluation scale.
Description of the aids set up within the framework of the personalized autonomy allowance for seniors program. | 90 days
  Formal home help can include several home services: meal delivery, domestic help, home care nurse, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, Haut-Rhin, France

IPD SHARING:
Plan to Share IPD: No